CLINICAL TRIAL: NCT01529411
Title: Randomized Phase II Study of Vinflunine as Maintenance Monotherapy in Patients With Advanced or Metastatic Urothelial Cancer That Obtains Clinical Benefit of the First Line With Cisplatin-gemcitabine Combination
Brief Title: Clinical Trial With Vinflunine as Maintenance Therapy in Metastatic Urothelial Cancer
Acronym: MAJA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Oncology Genito-Urinary Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOGUG2011/02
Record Dates: First submitted 2012-01-20; First posted 2012-02-08 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2012-02

CONDITIONS: Carcinoma, Transitional Cell
Keywords: urothelium; transitional; carcinoma; cancer; metastatic; tract
MeSH Terms: conditions — Carcinoma, Transitional Cell; Carcinoma; Neoplasms; Neoplasm Metastasis | interventions — vinflunine; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vinflunine (Experimental): Vinflunine 320 mg/m2 IV infusion in 20 minutes every 21 days (280mg/m2 if PS=1, age ≥ 75 years, previous pelvic radiotherapy or creatinine clearance < 60ml/min)
  + best suportive care, with regards clinical practice.
  Interventions: Drug: Vinflunine
- Best suportive care (Other): Best suportive care
  Interventions: Other: Undefined (standard care)

INTERVENTIONS:
Drug: Vinflunine — Vinflunine 320 mg/m2 IV infusion in 20 minutes every 21 days (280mg/m2 if PS=1, age ≥ 75 years, previous pelvic radiotherapy or creatinine clearance < 60ml/min).
  Other Names: Javlor
  Arms: Vinflunine
Other: Undefined (standard care) — All the current interventions used by each institution for the study disease.
  Other Names: undefined
  Arms: Best suportive care

SUMMARY:
This is a clinical trial to evaluate the efficacy and safety of the drug vinflunine administered after the standard treatment of the combination gemcitabine+cisplatin, when it has reached stabilization or response of the disease, as the first treatment inmeditely after the diagnosis of advanced or metastatic urothelial cancer.

DETAILED DESCRIPTION:
Vinflunine is a drug recently approved in Europe for the treatment of advanced or metastatic urothelial cancer after platinum-failure. It has proved to improve the survival results compared with the best suportive care. In adition, the tolerability was favourable, specially for not leading appearance of neuropathy nor other cumulative toxic effects.

In this study, it is proposed to test the feasibility, in terms of tolerability and efficacy of monotherapy with vinflunine in patients who, after completing the first-line cisplatin-based treatment for Transitional Cell Carcinoma of the Urothelial Tract (CCTU), have reached a stabilization or objective response. In order to have an adequate control group in the proposed design will be a phase II trial in which one group will receive standard management (follow-up until progression disease).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 & < 80
* Written informed consent given by the patient
* Diagnosis of urothelium cells transition cancer subsidiary locally advanced or metastatic resection
* One measurable target lesion minimum
* ECOG 0 or 1
* Stabilization or objective response after first-line treatment 6 cycles of cisplatin+gemcitabine
* Last administration of cisplatin and gemcitabine < 6 weeks
* Maximum grade I toxicity
* Adequate functions of bone marrow, kidney and liver
* Absence psychological, family, sociological or geographical disorder or other condition
* Women of childbearing potential must be using a medically accepted method of contraception (i.e. oral contraceptives, intrauterine devices) to avoid pregnancy during the 2 months preceding the start of study treatment, throughout the study period and for up to 3 months after the last dose of study treatment in such a manner that the risk of pregnancy is minimised. Women of childbearing potential must have a negative serum or urine pregnancy test within 72 hours prior to the start of study treatment.
* Fertile men must be using an effective method of birth control if their partners are women of childbearing potential up to 3 months after last administration of study medication.

Exclusion Criteria:

* ECOG > 2
* Patients with age > 80
* Patients with small cell carcinoma histology, lymphomas or sarcomas of the bladder.
* The patients that have received 7 or more cycles of a combination of cisplatin and gemcitabine in first line metastatic disease.
* Pregnant or lactating women or women with positive pregnancy test at screening, fertile sexual active women that did not use or do not wish or are unable to use an accepted method to prevent pregnancy during the 2 months prior to study treatment, during the study period and up to 3 months after the last dose of study treatment. Sexual active men who do not wish to use a method of birth during the study and up to 6 months after the last dose of study treatment if their partners are women of childbearing age.
* Known brain metastases or meningeal involvement. CT Scan not required to rule this unless there is clinical suspicion of disease of the central nervous system.
* Peripheral neuropathy grade 2 according to NCI-CTC version 4.0 [Common Toxicity Criteria of the National Cancer Institute].
* Prior radiation to > 30% of the bone marrow, radiation completed at least 30 days or current persistence of any adverse event.
* Other serious diseases or medical conditions like: systemic infection that required a systemic anti-infective treatment(grades 3 or 4 of the Common Toxicity Criteria NCI, version 4.03) and uncontrolled medical disorder, for example: patients with unstable angina or myocardial infarction within 6 months before registration or uncontrolled diabetes.
* Progressive Disease during 1st line treatment of advanced or metastatic disease with chemotherapy systemic cisplatin and gemcitabine.
* Patients who have received more than one line of treatment for metastatic disease.
* Patients who received cisplatin in monotherapy or in combination as neoadjuvant treatment, adjuvant after initial surgery of urothelial cancer.
* Patients treated with another investigational drug or treatment antineoplastic agent cisplatin or gemcitabine than within 30 days before randomization.
* Other cancers except basal skin cancer treated in an appropriate, cervical cancer in situ or other tumor a disease-free interval of 5 years.
* Inadequate renal function defined by a calculated clearance serum creatinine < 40 ml/min (Cockcroft-Gault).
* Known hypersensitivity to drug study or similar chemical structure drugs.
* Patients who require treatment with ketoconazole, itraconazole, ritonavir, amprenavir, indinavir, rifampin or phenytoin (any potent inhibitor or inducer of CYP3A4).
* Any concurrent chronic immunotherapy or prior organic allograft.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2012-02; Primary Completion 2013-02 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival. | 1 year
  To evaluate the Progression Free Survival (PFS) with vinflunine in maintenance monotherapy in patients with advanced or metastatic CCTU that has reached stabilization or objective response after completing 6 cycles with the combination cisplatin-gemcitabine in 1st line.

CONTACTS AND LOCATIONS:
Overall Officials: Jesús García-Donas, MD, Principal Investigator — Hospital Universitario Fundación Alcorcón; Albert Font, MD, Principal Investigator — ICO-Hospital Universitari Germans Trias i Pujol; Joaquim Bellmunt, MD, Principal Investigator — H. del Mar - FIMIM (Fundació Institut Mar d´Investigacions Mèdiques)
Locations (20):
- Spain (20):
  - Hospital General de Elda Virgen de la Salud, Elda, Alicante
  - ICO-Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - ICO-Hospital Duran i Reynals, L'Hospitalet de Llobregat, Barcelona
  - Hospital Fundació Althaia, Manresa, Barcelona
  - Corporació Sanitaria Parc Taulí, Sabadell, Barcelona
  - Complejo Hosp. Univ. de Santiago de Compostela, Santiago de Compostela, Galicia
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - H. del Mar (Fundació Institut Mar d´Investigacions Mèdiques - FIMIM), Barcelona
  - H. Universitari Vall d'Hebrón, Barcelona
  - Hospital Clínic i Provincial de Barcelona, Barcelona
  - H. General Universitario de Ciudad Real, Ciudad Real
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitari Son Espases, Palma de Mallorca
  - Clínica Universitaria de Navarra (CUN), Pamplona
  - Complejo Hospitalario de Navarra, Pamplona
  - H. Universitario Virgen de la Macarena, Seville
  - H. Universitario Virgen del Rocío, Seville
  - IVO, Valencia

REFERENCES:
- [Derived] Garcia-Donas J, Font A, Perez-Valderrama B, Virizuela JA, Climent MA, Hernando-Polo S, Arranz JA, Del Mar Llorente M, Lainez N, Villa-Guzman JC, Mellado B, Gonzalez Del Alba A, Castellano D, Gallardo E, Anido U, Garcia Del Muro X, Domenech M, Puente J, Morales-Barrera R, Perez-Gracia JL, Bellmunt J. Maintenance therapy with vinflunine plus best supportive care versus best supportive care alone in patients with advanced urothelial carcinoma with a response after first-line chemotherapy (MAJA; SOGUG 2011/02): a multicentre, randomised, controlled, open-label, phase 2 trial. Lancet Oncol. 2017 May;18(5):672-681a. doi: 10.1016/S1470-2045(17)30242-5. Epub 2017 Apr 4. PMID 28389316
- See also: Sponsor´s web-site — http://www.sogug.es